CLINICAL TRIAL: NCT00220532
Title: A Randomised Placebo-Controlled Trial to Evaluate Interactions Between Riboflavin and Folate Intake and Genotype in Reducing Risk of Cervical Cancer
Brief Title: Folate and Protection Against Cervical Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: World Cancer Research Fund International (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STH 13608
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Cervical Cancer
Keywords: Randomised placebo controlled intervention trial; Folic acid; Riboflavin; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Folic Acid; Riboflavin

INTERVENTIONS:
Drug: Folic acid with riboflavin

SUMMARY:
This is a randomised double-blind placebo-controlled trial to see whether giving a low dose of the vitamins folic acid and riboflavin is beneficial to women who have very low grade abnormalities of the cervical cells.

DETAILED DESCRIPTION:
The overall aim of the study is to evaluate interactions between intakes of folic acid and riboflavin with a common polymorphism relevant to folate metabolism, in determining the risk of cervical cancer in women who carry high risk human papillomavirus.

We will test the following hypotheses:

Supplements of riboflavin and folic acid will increase the rate of regression of low grade cervical intra epithelial neoplasia (CIN1).

Effects of supplemental folic acid and riboflavin on CIN1 regression are modulated by a common polymorphism in the MTHFRC677T gene.

We will recruit women with biopsy-proven CIN1 and carrying high risk HPV infection, and randomise to a 12month intervention of 1.2mg folic acid and 5mg riboflavin or placebo. The primary outcome will be regression of biopsy-proven CIN1, and secondary outcomes will include measures of DNA stability.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-diagnosed CIN1 infection with oncogenic HPV

Exclusion Criteria:

Any other stage of cervical abnormality pregnant or planning a pregnancy diabetic taking B vitamin supplements taking anti-epileptic treatment taking methotrexate bleeding after intercourse abnormal GI function infection with chlamydia, HIV or other agent

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180
Dates: Start 2005-07; Study Completion 2007-05

PRIMARY OUTCOMES:
Rate of regression of CIN1 to normal over a 12 month intervention

SECONDARY OUTCOMES:
DNA strand breakage, in cervical cells
DNA hypomethylation, in cervical cells
Cervical cell folic acid
HPV persistence over 12 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hilary J Powers, PhD, Principal Investigator — Human Nutrition Unit, University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom